CLINICAL TRIAL: NCT00707239
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Comparative Study Of The Safety And Efficacy of 2 Doses Of Tigecycline Versus Imipenem/Cilastatin For The Treatment Of Subjects With Hospital-Acquired Pneumonia
Brief Title: Study Evaluating Safety and Efficacy of Tigecycline Versus Imipenem/Cilastatin Subjects With Hospital-Acquired Pneumonia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3074K6-2000; B1811004
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Results first posted 2012-07-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-06

CONDITIONS: Pneumonia, Bacterial
Keywords: Hospital-acquired pneumonia; Ventilator-associated pneumonia
MeSH Terms: conditions — Pneumonia, Bacterial; Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated | interventions — Tigecycline; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental)
  Interventions: Drug: tigecycline
- B (Experimental)
  Interventions: Drug: tigecycline
- C (Active Comparator)
  Interventions: Drug: imipenem/cilastatin

INTERVENTIONS:
Drug: tigecycline — An initial intravenous (IV) loading dose of 150 mg of tigecycline, followed by 75 mg of IV tigecycline approximately every 12 hours (q12h), for up to 14 consecutive days. Ceftazidime 2 g IV approximately every 8 hours, an aminoglycoside (tobramycin 7mg/kg daily or amikacin 20 mg/kg daily) and vancomycin placebo given at the start of therapy (unless it is known at baseline that the subject does not have Pseudomonas aeruginosa or methicillin-resistant Staphylococcus aureus [MRSA]).
  Arms: A
Drug: tigecycline — An initial intravenous (IV) loading dose of 200 mg of tigecycline, followed by 100 mg of IV tigecycline approximately every 12 hours (q12h), for up to 14 consecutive days. Ceftazidime 2 g IV approximately every 8 hours, an aminoglycoside (tobramycin 7mg/kg daily or amikacin 20 mg/kg daily) and vancomycin placebo given at the start of therapy (unless it is known at baseline that the subject does not have Pseudomonas aeruginosa or methicillin-resistant Staphylococcus aureus [MRSA]).
  Arms: B
Drug: imipenem/cilastatin — Imipenem/cilastatin 1g intravenous (IV) will be administered approximately every 8 hours, for up to 14 consecutive days. In addition vancomycin 15 mg/kg IV approximately every 12 hours (q12h), an aminoglycoside (tobramycin 7mg/kg daily or amikacin 20 mg/kg daily) and ceftazidime placebo will be given at the start of therapy (unless it is known at baseline that the subject does not have Pseudomonas aeruginosa or methicillin-resistant Staphylococcus aureus [MRSA]).
  Arms: C

SUMMARY:
This study will compare the safety and efficacy of a tigecycline regimen versus an imipenem/cilastatin regimen for the treatment of subjects who are hospitalized with hospital-acquired pneumonia (HAP). At least 70% of enrolled subjects will have ventilator-associated pneumonia (VAP). Two dose levels of tigecycline will be assessed and compared to imipenem/cilastatin in parallel. Subjects will receive intravenous therapy from a minimum of 7 & up to 14 consecutive days, the exact duration will be at the decision of the investigator based on the subject's condition. Additional protocol specified antibiotics may be given to ensure appropriate coverage. A final assessment at test-of-cure (TOC) visit will be done 10 to 21 days after the last day of therapy. The total duration of subject participation will be between 17 and 44 days, including a follow up period of 30 days after the last day of therapy for SAEs.

Subjects will be followed for safety and efficacy. The safety assessment will include: physical examinations, vital signs, assessment of the clinical signs and symptoms of pneumonia, collection of adverse events, 12-lead ECG, collection of samples for hematology, serum chemistries, and coagulation parameters, & a serum or urine pregnancy test before study entry for women of childbearing potential. The clinical and microbiological efficacy will both be evaluated.

DETAILED DESCRIPTION:
The sponsor internal decision has been taken to close the study on 15 of July 2011, due to difficulties in enrollment. This decision was not based on any safety issues.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, greater than or equal to 18 years of age, known or suspected to have acute hospital-acquired pneumonia (HAP).
* Acute HAP is defined as pneumonia with onset of symptoms:

  1. Greater than or equal to 48 hours after admission to an acute care hospital or chronic care facility such as a skilled nursing home facility or rehabilitation unit. Or
  2. Less than or equal to 7 days after the subject was discharged from the hospital. The initial hospitalization must have been greater than or equal to 3 days duration.
* VAP is defined as: onset of symptoms of pneumonia greater than or equal to 48 hours after endotracheal intubation.
* Presence of a new or evolving infiltrate on a chest x-ray film, presence of fever or leukocytosis, respiratory failure requiring mechanical ventilation or presence of 2 of the following clinical signs and symptoms: cough, dyspnea or tachypnea, pleuritic chest pain, rales and/or evidence of pulmonary consolidation, hypoxemia, or purulent sputum production.

Exclusion Criteria:

* Subjects with other significant underlying conditions that would make it difficult to evaluate the subjects or make it unlikely to complete the therapy or that would increase their risk by participating in the study, infection with organisms known to be resistant, contraindication, or hypersensitivity to any of the test articles.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- United States (3):
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Morgantown, West Virginia
- Argentina (3):
  - Pfizer Investigational Site, La Plata, Buenos Aires
  - Pfizer Investigational Site, Godoy Cruz, Mendoza Province
  - Pfizer Investigational Site, Provincia de Buenos Aires
- Australia (2):
  - Pfizer Investigational Site, Nambour, Queensland
  - Pfizer Investigational Site, Victoria, Victoria
- Brazil (3):
  - Pfizer Investigational Site, Belo Horizonte, Minas Gerais
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São José do Rio Preto, São Paulo
- Canada (2):
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Trois-Rivières, Quebec
- Pfizer Investigational Site, Santiago, Santiago Metropolitan, Chile
- Colombia (2):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Bogotá
- Pfizer Investigational Site, Zagreb, Croatia
- Pfizer Investigational Site, Argenteuil, France
- Hungary (4):
  - Pfizer Investigational Site, Debrecen
  - Pfizer Investigational Site, Nyíregyháza
  - Pfizer Investigational Site, Székesfehérvár
  - Pfizer Investigational Site, Vác
- Latvia (2):
  - Pfizer Investigational Site, Daugavpils
  - Pfizer Investigational Site, Riga
- Russia (4):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Novosibirsk
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Vsevolozhsk
- Pfizer Investigational Site, Seoul, Korea, South Korea
- Taiwan (4):
  - Pfizer Investigational Site, Tainan, Taiwan
  - Pfizer Investigational Site, Taipei, Taiwan
  - Pfizer Investigational Site, Tainan
  - Pfizer Investigational Site, Taipei TOC

REFERENCES:
- [Derived] Ramirez J, Dartois N, Gandjini H, Yan JL, Korth-Bradley J, McGovern PC. Randomized phase 2 trial to evaluate the clinical efficacy of two high-dosage tigecycline regimens versus imipenem-cilastatin for treatment of hospital-acquired pneumonia. Antimicrob Agents Chemother. 2013 Apr;57(4):1756-62. doi: 10.1128/AAC.01232-12. Epub 2013 Jan 28. PMID 23357775
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3074K6-2000&StudyName=Study%20Evaluating%20Safety%20and%20Efficacy%20of%20Tigecycline%20Versus%20Imipenem/Cilastatin%20Subjects%20With%20Hospital-Acquired%20Pneumonia

RESULTS

PARTICIPANT FLOW:
Groups:
- Tigecycline 75 mg: Tigecycline 150 milligram (mg) loading dose intravenously followed by tigecycline 75 mg maintenance dose intravenously approximately every 12 hours (hrs). Ceftazidime 2 gram intravenously approximately every 8 hrs, an aminoglycoside (tobramycin 7 mg/kilogram [mg/kg] or amikacin 20 mg/kg daily) and vancomycin placebo intravenously at the start of therapy unless participant did not have Pseudomonas aeruginosa (P. aeruginosa) or methicillin-resistant Staphylococcus aureus (MRSA).
- Tigecycline 100 mg: Tigecycline 200 mg loading dose intravenously followed by tigecycline 100 mg maintenance dose intravenously approximately every 12 hrs. Ceftazidime 2 gram intravenously approximately every 8 hrs, an aminoglycoside (tobramycin 7 mg/kg or amikacin 20 mg/kg daily) and vancomycin placebo intravenously at the start of therapy unless participant did not have P. aeruginosa or MRSA.
- Imipenem/Cilastatin 1 Gram: Imipenem/cilastatin 1 gram intravenously approximately every 8 hrs. Vancomycin 15 mg/kg intravenously approximately every 12 hrs, an aminoglycoside (tobramycin 7 mg/kg or amikacin 20 mg/kg daily) and ceftazidime placebo intravenously at the start of therapy unless participant did not have P. aeruginosa or MRSA.
Period: Overall Study
Arm/Group | Tigecycline 75 mg | Tigecycline 100 mg | Imipenem/Cilastatin 1 Gram
Started | 37 | 36 | 35
Treated | 36 | 35 | 34
Completed | 18 | 25 | 21
Not Completed | 19 | 11 | 14
Not completed — Adverse Event | 5 | 3 | 2
Not completed — Death | 3 | 1 | 3
Not completed — Physician Decision | 1 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 2 | 0
Not completed — Randomized, but not treated | 1 | 1 | 1
Not completed — Other | 8 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tigecycline 75 mg | Tigecycline 100 mg | Imipenem/Cilastatin 1 Gram | Total
Number analyzed (Participants) | 36 | 35 | 34 | 105
Age Continuous [Mean (Standard Deviation); unit: years] | 60.31 (14.82) | 61.46 (16.05) | 64.85 (15.33) | 62.16 (15.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 5 | 34
  Male | 23 | 19 | 29 | 71

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Response in Clinically Evaluable (CE) Population at Test-of-Cure (TOC) Visit
Description: Clinical response: Cure=All initial signs/symptoms of pneumonia (SSx) improved; chest x-ray (CXR) improved/stable; no other antibiotics for pneumonia; no worsening or new SSx. Failure=Persistence or worsening SSx; no clinical improvement or initial improvement with clinically important worsening; other antimicrobials for pneumonia; CXR progression; death > study day 2 due to pneumonia. Indeterminate=unable to determine outcome for non-study drug/infection reasons (e.g., lost to follow-up); death in 2 days after 1st dose for any reason, or >2 days but before TOC visit for non-pneumonia reason.
Time Frame: Up to Day 24 to 35 (10 to 21 days after last day of therapy [LDOT])
Population: CE population included those participants who met specified evaluability criteria for efficacy.
Measure: Number; unit: percentage of participants
Arm/Group | Tigecycline 75 mg | Tigecycline 100 mg | Imipenem/Cilastatin 1 Gram
Number analyzed (Participants) | 23 | 20 | 24
percentage of participants
  Cure | 69.6 | 85.0 | 75.0
  Failure | 30.4 | 15.0 | 25.0
Statistical Analysis 1: Comparison: Tigecycline 75 mg vs Imipenem/Cilastatin 1 Gram; Cure: Confidence interval (CI) was calculated using the Wilson score method, with continuity correction. Clinical response (rates of cure) by using a 2-sided 70 percent (%) CI for the true difference in efficacy (tigecycline regimen minus imipenem/cilastatin regimen) was calculated. Statistical testing was done at 15% alpha; Test type: Superiority or Other; Risk Difference (RD) = -5.4, 70% CI 2-sided [-21.6 to 10.9]
Statistical Analysis 2: Comparison: Tigecycline 100 mg vs Imipenem/Cilastatin 1 Gram; Cure: CI was calculated using the Wilson score method, with continuity correction. Clinical response (rates of cure) by using a 2-sided 70% CI for the true difference in efficacy (tigecycline regimen minus imipenem/cilastatin regimen) was calculated. Statistical testing was done at 15% alpha; Test type: Superiority or Other; Risk Difference (RD) = 10.0, 70% CI 2-sided [-6.1 to 24.8]

2. Secondary Outcome: Percentage of Participants With Clinical Response in Clinical Modified Intent-to-treat (c-mITT) Population at Test-of-Cure (TOC) Visit
Description: Clinical response: Cure=All initial SSx improved; CXR improved/stable; no other antibiotics for pneumonia; no worsening or new SSx. Failure=Persistence or worsening SSx; no clinical improvement or initial improvement with clinically important worsening; other antimicrobials for pneumonia; CXR progression; death > study day 2 due to pneumonia. Indeterminate=unable to determine outcome for non-study drug/infection reasons (e.g., lost to follow-up); death in 2 days after 1st dose for any reason, or >2 days but before TOC visit for non-pneumonia reason.
Time Frame: Up to Day 24 to 35 (10 to 21 days after LDOT)
Population: c-mITT population included all participants who were randomly assigned to receive intravenous study medication and had clinical evidence of hospital-acquired pneumonia (HAP).
Measure: Number; unit: percentage of participants
Arm/Group | Tigecycline 75 mg | Tigecycline 100 mg | Imipenem/Cilastatin 1 Gram
Number analyzed (Participants) | 36 | 35 | 34
percentage of participants
  Cure | 52.8 | 71.4 | 52.9
  Failure | 27.8 | 14.3 | 17.6
  Indeterminate | 19.4 | 14.3 | 29.4
Statistical Analysis 1: Comparison: Tigecycline 75 mg vs Imipenem/Cilastatin 1 Gram; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Risk Difference (RD) = -0.2, 70% CI 2-sided [-14.3 to 14.0]
Statistical Analysis 2: Comparison: Tigecycline 100 mg vs Imipenem/Cilastatin 1 Gram; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Risk Difference (RD) = 18.5, 70% CI 2-sided [4.3 to 31.8]

3. Secondary Outcome: Percentage of Participants With Clinical Response in Ventilator Associated Pneumonia (VAP) and Non-VAP Participants at Test-of-Cure (TOC) Visit
Description: as for outcome 2
Time Frame: Up to Day 24 to 35 (10 to 21 days after LDOT)
Population: CE population included those participants who met specified evaluability criteria for efficacy. 'n' is signifying those participants who were evaluable for this measure and included in VAP (suffering from VAP) and non-VAP group (not suffering from VAP) for each group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Tigecycline 75 mg | Tigecycline 100 mg | Imipenem/Cilastatin 1 Gram
Number analyzed (Participants) | 23 | 20 | 24
percentage of participants
  VAP: Cure (n = 7, 7, 9) | 71.4 | 85.7 | 77.8
  VAP: Failure (n = 7, 7, 9) | 28.6 | 14.3 | 22.2
  Non-VAP: Cure (n = 16, 13, 15) | 68.8 | 84.6 | 73.3
  Non-VAP: Failure (n = 16, 13, 15) | 31.3 | 15.4 | 26.7

4. Secondary Outcome: Percentage of Participants With Microbiological Response at the Pathogen Level Population at Test-of-Cure (TOC) Visit
Description: Eradication=baseline isolate not present in repeat culture from the original infection site; Presumed Eradication=clinical response of cure precluded the availability of a specimen for culture; Persistence=baseline isolate present in repeat culture from the original infection site; Presumed Persistence=culture data not available for participants with a clinical response of failure; Indeterminate=unable to determine outcome for non-study drug/infection reasons; no baseline isolate; death in 2 days after 1st dose for any reason, or >2 days but before TOC visit for non-pneumonia reason.
Time Frame: Up to Day 24 to 35 (10 to 21 days after LDOT)
Population: Microbiologically Evaluable (ME) population:participants who met evaluability criteria for efficacy, had culture taken from infected site before dose 1 of study drug, had at least (>=)1 pathogen, >=1 pathogen was susceptible to tigecycline, imipenem/cilastatin regimen; 'n' = those participants who had specified pathogen for each group respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Tigecycline 75 mg | Tigecycline 100 mg | Imipenem/Cilastatin 1 Gram
Number analyzed (Participants) | 13 | 10 | 15
percentage of participants
  Acinetobacter calcoaceticus: Eradication (n=3,2,3) | 66.7 | 50.0 | 66.7
  Acinetobacter calcoaceticus: Persistence (n=3,2,3) | 33.3 | 50.0 | 33.3
  Enterobacter cloacae: Eradication (n=0,0,2) | NA — Data was not available since none of the participants in this reporting group were affected with Enterobacter cloacae. | NA — Data was not available since none of the participants in this reporting group were affected with Enterobacter cloacae. | 50.0
  Enterobacter cloacae: Persistence (n=0,0,2) | NA — Data was not available since none of the participants in this reporting group were affected with Enterobacter cloacae. | NA — Data was not available since none of the participants in this reporting group were affected with Enterobacter cloacae. | 50.0
  Escherichia coli: Eradication (n=1,1,2) | 0 | 0 | 50.0
  Escherichia coli: Persistence (n=1,1,2) | 100.0 | 100.0 | 50.0
  Haemophilus: Eradication (n=1,0,0) | 100.0 | NA — Data was not available since none of the participants in this reporting group were affected with Haemophilus. | NA — Data was not available since none of the participants in this reporting group were affected with Haemophilus.
  Haemophilus influenzae: Eradication (n=0,1,1) | NA — Data was not available since none of the participants in this reporting group were affected with Haemophilus influenzae. | 100.0 | 0
  Haemophilus influenzae: Persistence (n=0,1,1) | NA — Data was not available since none of the participants in this reporting group were affected with Haemophilus influenzae. | 0 | 100.0
  Klebsiella oxytoca: Eradication (n=1,0,0) | 100.0 | NA — Data was not available since none of the participants in this reporting group were affected with Klebsiella oxytoca. | NA — Data was not available since none of the participants in this reporting group were affected with Klebsiella oxytoca.
  Klebsiella pneumoniae: Eradication (n=2,2,5) | 50.0 | 50.0 | 80.0
  Klebsiella pneumoniae: Persistence (n=2,2,5) | 50.0 | 50.0 | 20.0
  Serratia marcescens: Eradication (n=0,2,0) | NA — Data was not available since none of the participants in this reporting group were affected with Serratia marcescens. | 100.0 | NA — Data was not available since none of the participants in this reporting group were affected with Serratia marcescens.
  Staphylococcus aureus (SA): Eradication (n=8,6,9) | 62.5 | 83.3 | 88.9
  SA: Persistence (n=8,6,9) | 37.5 | 16.7 | 11.1
  MRSA:Eradication (n=4,2,4) | 50.0 | 100.0 | 100.0
  MRSA:Persistence (n=4,2,4) | 50.0 | 0 | 0
  Methicillin-suseptible SA: Eradication (n=4,4,5) | 75.0 | 75.0 | 80.0
  Methicillin-suseptible SA: Persistence (n=4,4,5) | 25.0 | 25.0 | 20.0
  Streptococcus anginosus: Eradication (n=1,0,0) | 100.0 | NA — Data was not available since none of the participants in this reporting group were affected with Streptococcus anginosus. | NA — Data was not available since none of the participants in this reporting group were affected with Streptococcus anginosus.
  Streptococcus mitis: Eradication (n=1,0,0) | 100.0 | NA — Data was not available since none of the participants in this reporting group were affected with Streptococcus mitis. | NA — Data was not available since none of the participants in this reporting group were affected with Streptococcus mitis.
  Streptococcus oralis: Eradication (n=0,0,1) | NA — Data was not available since none of the participants in this reporting group were affected with Streptococcus oralis. | NA — Data was not available since none of the participants in this reporting group were affected with Streptococcus oralis. | 100.0
  Streptococcus pneumonia: Eradication (n=1,1,0) | 100.0 | 100.0 | NA — Data was not available since none of the participants in this reporting group were affected with Streptococcus pneumonia.

5. Secondary Outcome: Percentage of Participants With Microbiological Response at the Participant Level Population at Test-of-Cure (TOC) Visit
Description: Microbiological response assessed at participant level. Eradication = baseline isolate not present in repeat culture from the original infection site; Presumed Eradication = clinical response of cure precluded the availability of a specimen for culture; Persistence = baseline isolate present in repeat culture from the original infection site; Presumed Persistence = culture data not available for participants with a clinical response of failure; Superinfection = culture from the primary infection site had new pathogen not identified as a baseline isolate and clinical response was failure.
Time Frame: Up to Day 24 to 35 (10 to 21 days after LDOT)
Population: ME population included participants who met specified evaluability criteria for efficacy, had culture taken from the infected site before first dose of study medication and had at least 1 pathogen, and at least 1 baseline pathogen was susceptible to tigecycline and imipenem/cilastatin regimens.
Measure: Number; unit: percentage of participants
Arm/Group | Tigecycline 75 mg | Tigecycline 100 mg | Imipenem/Cilastatin 1 Gram
Number analyzed (Participants) | 13 | 10 | 15
percentage of participants
  Eradication | 61.5 | 80.0 | 80.0
  Persistence | 38.5 | 20.0 | 13.3
  Superinfection | 0.0 | 0.0 | 6.7
Statistical Analysis 1: Comparison: Tigecycline 75 mg vs Imipenem/Cilastatin 1 Gram; Eradication: CI was calculated using the Wilson score method, with continuity correction. Microbiological response (rates of eradication) by using a 2-sided 70% CI for the true difference in efficacy (tigecycline regimen minus imipenem/cilastatin regimen) was calculated. Statistical testing was done at 15% alpha; Test type: Superiority or Other; Risk Difference (RD) = -18.5, 70% CI 2-sided [-39.6 to 4.2]
Statistical Analysis 2: Comparison: Tigecycline 100 mg vs Imipenem/Cilastatin 1 Gram; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; Risk Difference (RD) = 0.0, 70% CI 2-sided [-23.8 to 20.9]

6. Other Pre Specified Outcome: Number of Participants Who Experienced Nausea or Vomiting
Time Frame: Baseline up to Day 29 to Day 35 (15 to 21 days after LDOT)
Population: Modified intent-to-treat (mITT) population included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Tigecycline 75 mg | Tigecycline 100 mg | Imipenem/Cilastatin 1 Gram
Number analyzed (Participants) | 36 | 35 | 34
participants
  Nausea | 1 | 3 | 1
  Vomiting | 3 | 1 | 4
Statistical Analysis 1: Comparison: Tigecycline 75 mg vs Tigecycline 100 mg vs Imipenem/Cilastatin 1 Gram; Nausea: p-value was calculated using 2-tail Fischer's exact test; Test type: Superiority or Other; p = 0.527, Fisher Exact — Statistical testing was done at 5% alpha
Statistical Analysis 2: Comparison: Tigecycline 75 mg vs Tigecycline 100 mg vs Imipenem/Cilastatin 1 Gram; Vomiting: p-value was calculated using 2-tail Fischer's exact test; Test type: Superiority or Other; p = 0.390, Fisher Exact — Statistical testing was done at 5% alpha

7. Other Pre Specified Outcome: Number of Participants With Abnormal Laboratory Examinations
Description: Participants were evaluated for following laboratory parameters: albumin, alkaline phosphatase, amylase, urea (blood urea nitrogen [BUN]), total bilirubin, calcium, magnesium, carbon dioxide, international normalized ratio (INR), chloride, creatinine, glucose, lipase, potassium, phosphorus, aspartate aminotransferase (AST), alanine aminotransferase (ALT), sodium, total protein, hemoglobin, hematocrit, white blood cells, eosinophils, neutrophils, lymphocytes, platelets, prothrombin time, prothrombin activity and partial thromboplastin time.
Time Frame: Baseline up to Day 24 to Day 35 (10 to 21 days after LDOT)
Population: mITT population included all randomized participants who received at least 1 dose of study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | Tigecycline 75 mg | Tigecycline 100 mg | Imipenem/Cilastatin 1 Gram
Number analyzed (Participants) | 36 | 33 | 33
participants | 34 | 31 | 31
Statistical Analysis 1: Comparison: Tigecycline 75 mg vs Tigecycline 100 mg vs Imipenem/Cilastatin 1 Gram; p-value was calculated using 2-tail Fischer's exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact — Statistical testing was done at 5% alpha

8. Other Pre Specified Outcome: Number of Participants With Abnormal Electrocardiogram (ECG)
Description: Potentially clinically significant ECG data: Non-first values greater than 240 millisecond (msec) with increase of greater than or equal to 10 percent (%) from baseline for PR interval; Non-first values greater than or equal to 120 msec for QRS interval; Non-first values greater than 460 msec with increase of greater than or equal to 5% from baseline for corrected QT (QTc) interval; Non-first values greater than 460 msec with increase of greater than or equal to 5% from baseline for QTc using Framingham formula (QTc F).
Time Frame: Baseline up to Day 14 or LDOT
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Tigecycline 75 mg | Tigecycline 100 mg | Imipenem/Cilastatin 1 Gram
Number analyzed (Participants) | 35 | 33 | 33
participants | 14 | 14 | 14
Statistical Analysis 1: Comparison: Tigecycline 75 mg vs Tigecycline 100 mg vs Imipenem/Cilastatin 1 Gram; p-value was calculated using 2-tail Fischer's exact test; Test type: Superiority or Other; p = 1.000, Fisher Exact — Statistical testing was done at 5% alpha

9. Other Pre Specified Outcome: Maximum Observed Serum Concentration (Cmax) of Tigecycline
Time Frame: Day 3, 4 or 5
Population: CE population included those participants who met specified evaluability criteria for efficacy. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Tigecycline 75 mg | Tigecycline 100 mg
Number analyzed (Participants) | 20 | 19
nanogram/milliliter (ng/mL) | 479 (327) | 1217 (1070)

10. Other Pre Specified Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of Tigecycline
Time Frame: Day 3, 4 or 5
Population: as for outcome 9
Measure: Median (Full Range); unit: hrs
Arm/Group | Tigecycline 75 mg | Tigecycline 100 mg
Number analyzed (Participants) | 20 | 19
hrs | 0.5 [0.5 to 8.0] | 0.5 [0.5 to 2.0]

11. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-12)] of Tigecycline
Description: AUC (0-12) = Area under the serum concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-12). Area under the serum concentration-time curve was derived from the population pharmacokinetic (PK) analysis by using each participant's dose and the post-hoc individual estimated systemic CL, AUC (0-12) = Dose divided by CL.
Time Frame: Day 3, 4 or 5
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Tigecycline 75 mg | Tigecycline 100 mg
Number analyzed (Participants) | 20 | 19
ng*hr/mL | 3.20 (1.28) | 5.04 (1.31)

12. Other Pre Specified Outcome: Clearance (CL) of Tigecycline
Description: Drug clearance (CL) is a quantitative measure of the rate at which a drug substance is removed from the blood. It is defined as the volume of serum from which drug can be completely removed per unit of time.
Time Frame: Day 3, 4 or 5
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: Liter/hr
Groups:
- Tigecycline: Tigecycline 150 or 200 mg loading dose intravenously followed by tigecycline 75 or 100 mg maintenance dose intravenously approximately every 12 hrs. Ceftazidime 2 gram intravenously approximately every 8 hrs, an aminoglycoside (tobramycin 7 mg/kg or amikacin 20 mg/kg daily) and vancomycin placebo intravenously at the start of therapy unless the participant did not have P. aeruginosa or MRSA.
Arm/Group | Tigecycline
Number analyzed (Participants) | 39
Liter/hr | 22.6 [19.4 to 26.4]

13. Other Pre Specified Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-24)] of Tigecycline
Description: AUC (0-24) = Area under the serum concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-24). Area under the serum concentration-time curve was derived from the population pharmacokinetic (PK) analysis by using each participant's dose and the post-hoc individual estimated systemic CL, AUC (0-12) = Dose divided by CL. Model-predicted AUC (0-24) was calculated by multiplying AUC (0-12) by 2.
Time Frame: Day 3, 4 or 5
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg*hr/mL
Arm/Group | Tigecycline 75 mg | Tigecycline 100 mg
Number analyzed (Participants) | 20 | 19
mg*hr/mL | 6.40 (2.55) | 10.07 (2.61)

14. Other Pre Specified Outcome: Correlation of AUC (0-24) of Tigecycline With Nausea and Vomiting
Description: AUC (0-24) = Area under the serum concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-24). Area under the serum concentration-time curve was derived from the population PK analysis by using each participant's dose and the post-hoc individual estimated systemic CL, AUC (0-12) = Dose divided by CL. Model-predicted AUC (0-24) was calculated by multiplying AUC (0-12) by 2.
Time Frame: Baseline up to Day 29 to 35 (15 to 21 days after LDOT)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg*hr/mL
Arm/Group | Tigecycline
Number analyzed (Participants) | 39
mg*hr/mL
  Experienced nausea (n = 4) | 8.668 (4.401)
  Did not experience nausea (n = 35) | 8.206 (3.102)
  Experienced vomiting (n = 4) | 6.863 (3.065)
  Did not experience vomiting (n = 35) | 8.412 (3.205)
Statistical Analysis 1: Comparison: Tigecycline; Statistical analysis was carried out between categories, experienced nausea and did not experience nausea; Test type: Superiority or Other; p = 0.78, Regression, Logistic; Odds Ratio (OR) = 1.0479, 95% CI 2-sided [0.754 to 1.46]
Statistical Analysis 2: Comparison: Tigecycline; Statistical analysis was carried out between categories, experienced vomiting and did not experience vomiting; Test type: Superiority or Other; p = 0.356, Regression, Logistic; Odds Ratio (OR) = 0.84644, 95% CI 2-sided [0.593 to 1.21]

15. Other Pre Specified Outcome: Correlation of AUC(0-24) to Minimum Inhibitory Concentration (MIC) Ratio (AUC [0-24]/MIC) of Tigecycline With Clinical Outcome
Description: Clinical response:Cure =Initial SSx improved;CXR improved/stable;no other antibiotic for pneumonia;no worsening/new SSx. Failure=Persistence/worsening SSx;no clinical improvement/initial improvement with worsening; other antibiotic;CXR progression;death >study day 2 due to pneumonia. Indeterminate=unable to determine outcome for non-study drug/infection reason;death in 2 days after dose 1 for any reason or >2 days but before TOC visit for non-pneumonia reason. MIC=lowest drug concentration with no visible growth of microorganism. AUC(0-24)/MIC:reported for cure and failure/indeterminate.
Time Frame: Up to Day 24 to 35 (10 to 21 days after LDOT)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tigecycline
Number analyzed (Participants) | 25
ratio
  Cure (n = 17) | 24.3 (20.4)
  Failure/indeterminate (n = 8) | 22.8 (9.59)
Statistical Analysis 1: Comparison: Tigecycline; Statistical analysis was carried out between categories, cure and failure/indeterminate; Test type: Superiority or Other; p = 0.836, Regression, Logistic; Odds Ratio (OR) = 1.0054, 95% CI 2-sided [0.956 to 1.06]

16. Other Pre Specified Outcome: Correlation of AUC(0-24) to Minimum Inhibitory Concentration (MIC) Ratio (AUC [0-24]/MIC) of Tigecycline With Microbiological Outcome
Description: Microbiological response:Eradication=baseline isolate not present in repeat culture from original infection site;Presumed Eradication=clinical response of cure precluded availability of specimen for culture;Persistence=baseline isolate present in repeat culture from original infection site;Presumed Persistence=culture data not available for participants with clinical response of failure;Superinfection=culture from primary infection site had new pathogen not identified as baseline isolate, clinical response was failure. MIC=lowest drug concentration with no visible growth of microorganism.
Time Frame: Up to Day 24 to 35 (10 to 21 days after LDOT)
Population: Data was not analyzed because correlation analysis could not be performed due to insufficient number of participants for whom data for both microbiological outcomes and tigecycline concentration was available.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Tigecycline
Number analyzed (Participants) | 0

17. Other Pre Specified Outcome: Maximum Observed Plasma Concentration of Procalcitonin (Cmaxpd) and Predicted Procalcitonin Plasma Concentration at 24 Hours (Cpd,24) and 48 Hours (Cpd,48)
Time Frame: Baseline up to Day 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Tigecycline or Imipenem/Cilastatin: Tigecycline 150 or 200 mg loading dose intravenously followed by tigecycline 75 or 100 mg maintenance dose intravenously approximately every 12 hrs or imipenem/cilastatin 1 gram intravenously approximately every 8 hrs. Ceftazidime 2 gram or matching placebo intravenously approximately every 8 hrs, an aminoglycoside, either tobramycin 7 mg/kg daily or amikacin 20 mg/kg daily, and vancomycin 15 mg/kg or matching placebo intravenously at the start of therapy unless it was known at baseline that the participant did not have P. aeruginosa or MRSA.
Arm/Group | Tigecycline or Imipenem/Cilastatin
Number analyzed (Participants) | 98
ng/mL
  Cmax | 2.83 (8.29)
  Cpd,24 | 1.86 (4.54)
  Cpd,48 | 1.74 (4.12)

18. Other Pre Specified Outcome: Time to Reach Half of the Maximum Observed Plasma Concentration and Time to Normalization of Concentrations (Tnorm) of Procalcitonin
Time Frame: Baseline up to Day 6
Population: Data was not analyzed because there was no apparent change in procalcitonin concentration over time.
Measure: Median (Full Range); unit: hr
Groups:
- Tigecycline or Imipenem/Cilastatin: Tigecycline 150 or 200 mg loading dose intravenously followed by tigecycline 75 or 100 mg maintenance dose intravenously approximately every 12 hrs or imipenem/cilastatin 1 gram intravenously approximately every 8 hrs. Ceftazidime 2 gram or matching placebo intravenously approximately every 8 hrs, an aminoglycoside, either tobramycin 7 mg/kg daily or amikacin 20 mg/kg daily, and vancomycin 15 mg/kg or matching placebo intravenously every 12 hrs at the start of therapy unless it was known at baseline that the participant did not have P. aeruginosa or MRSA.
Arm/Group | Tigecycline or Imipenem/Cilastatin
Number analyzed (Participants) | 0

19. Other Pre Specified Outcome: Duration of Intravenous Antibiotic Treatment, Hospital and Intensive Care Unit (ICU) Stay
Time Frame: Baseline up to Day 44 (30 days after LDOT)
Population: mITT population included all randomized participants who received at least 1 dose of study medication. Here, 'n' signifies those participants who were evaluable for intravenous antibiotic treatment, hospital or ICU stay for each reporting group respectively.
Measure: Median (Full Range); unit: days
Arm/Group | Tigecycline 75 mg | Tigecycline 100 mg | Imipenem/Cilastatin 1 Gram
Number analyzed (Participants) | 36 | 35 | 34
days
  Intravenous antibiotic treatment (n = 36, 35, 34) | 8.00 [2.00 to 15.00] | 9.00 [1.00 to 15.00] | 8.50 [1.00 to 15.00]
  Hospital stay (n = 36, 35, 34) | 13.00 [2.00 to 29.00] | 13.00 [1.00 to 26.00] | 15.50 [2.00 to 32.00]
  ICU stay (n = 25, 25, 29) | 8.00 [2.00 to 16.00] | 9.00 [1.00 to 24.00] | 10.00 [2.00 to 25.00]
Statistical Analysis 1: Comparison: Tigecycline 75 mg vs Tigecycline 100 mg vs Imipenem/Cilastatin 1 Gram; Intravenous antibiotic treatment: One-way analysis of variance (ANOVA) with treatment as factor was used to calculate p-value; Test type: Superiority or Other; p = 0.245, ANOVA — Statistical testing was done at 5% alpha
Statistical Analysis 2: Comparison: Tigecycline 75 mg vs Tigecycline 100 mg vs Imipenem/Cilastatin 1 Gram; Hospital stay: One-way ANOVA with treatment as factor was used to calculate p-value; Test type: Superiority or Other; p = 0.484, ANOVA — Statistical testing was done at 5% alpha
Statistical Analysis 3: Comparison: Tigecycline 75 mg vs Tigecycline 100 mg vs Imipenem/Cilastatin 1 Gram; ICU stay: One-way ANOVA with treatment as factor was used to calculate p-value; Test type: Superiority or Other; p = 0.192, ANOVA — Statistical testing was done at 5% alpha

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tigecycline 75 mg | Tigecycline 100 mg | Imipenem/Cilastatin 1 Gram
Serious Adverse Events (participants affected / at risk) | 12/36 | 9/35 | 10/34
Other Adverse Events (participants affected / at risk) | 28/36 | 25/35 | 26/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tigecycline 75 mg (N=36) | Tigecycline 100 mg (N=35) | Imipenem/Cilastatin 1 Gram (N=34)
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 2
Sinoatrial block (Cardiac disorders) | 0 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
Candida sepsis (Infections and infestations) | 0 | 1 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Septic shock (Infections and infestations) | 4 | 1 | 2
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Tracheal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Vascular disorders (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Deep vein thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Shock (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tigecycline 75 mg (N=36) | Tigecycline 100 mg (N=35) | Imipenem/Cilastatin 1 Gram (N=34)
Activated partial thromboplastin time prolonged (Investigations) | 0 | 2 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 3 | 4 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 6
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Constipation (Gastrointestinal disorders) | 1 | 2 | 6
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 6 | 5
Hypertension (Vascular disorders) | 0 | 3 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 3 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 1 | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 2
Lipase increased (Investigations) | 3 | 3 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 4 | 1
Oedema peripheral (General disorders) | 2 | 0 | 1
Oxygen saturation decreased (Investigations) | 2 | 0 | 0
Pain (General disorders) | 0 | 0 | 2
Phlebitis (Vascular disorders) | 2 | 0 | 0
Postoperative wound infection (Infections and infestations) | 2 | 0 | 0
Pyrexia (General disorders) | 3 | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 4 | 2 | 4

LIMITATIONS AND CAVEATS:
Formal statistical conclusions could not be made due to premature termination of study, because of enrollment difficulties, and small number of enrolled participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.